CLINICAL TRIAL: NCT03470337
Title: Phlogenzym® in Patients With Acute Thrombophlebitis - Efficacy and Tolerance - Randomised Double-blind Study Phase III With Parallel Groups vs. Placebo According to the Guidelines of Good Clinical Practice (GCP)
Brief Title: Phlogenzym® in Patients With Acute Thrombophlebitis - Efficacy and Tolerance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mucos Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MU-696414
Record Dates: First submitted 2018-03-06; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Thrombophlebitis Leg
Keywords: Thrombophlebitis
MeSH Terms: conditions — Thrombophlebitis | interventions — Phlogenzym; Wobenzym

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phlogenzym (Experimental): Treatment with German licensed drug Phlogenzym (6 tablets/day)
  Interventions: Drug: Phlogenzym
- Placebo (Placebo Comparator): Placebo equates Phlogenzym but without active ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phlogenzym — Bromelain / Trypsin / Rutoside
  Other Names: Wobenzym plus
  Arms: Phlogenzym
Other: Placebo
  Arms: Placebo

SUMMARY:
Oral enzyme therapy in patients with acute superficial vein inflammation (thrombophlebitis) can serve as an additional treatment option besides standard therapy with compression stockings, common pain medication and physical treatments. This randomized, double-blinded trial compares efficacy and safety with placebo.

DETAILED DESCRIPTION:
Enzymes are absorbed in the small intestine and taken up into the bloodstream, at least to some extent. There, they act in an anti-inflammatory manner, as was first described for the serine protease trypsin. Similarly, the cysteine protease bromelain, extracted from the stems of pineapples, is an effective phytotherapeutical drug with anti-inflammatory properties.Proteases have also been indicated to show a certain improvement of the fluidity of the blood. An additional component of the oral enzyme combination can be rutoside, or rutin, a flavonoid known to have cytoprotective and anti-inflammatory properties.

ELIGIBILITY:
Inclusion Criteria:

* male ог female patients with thrombophlebitis in the upper extremities (with ог without varicosis);
* age ~ 18 years;
* acute thrombophlebitis in the lower leg
* moderate to severe pain as monitored on a visual analog scale (VAS, value ≥ 3 cm)
* pain under pressure
* presence of at least three of the following symptoms: skin redness, hyperthermia, phlebitic cords, feeling of heaviness and tenseness.

Exclusion Criteria:

* known deep phlebothrombosis
* flourishing ulcus cruris
* arterial occlusive disease
* peripheral neuropathy
* malignant disease
* concomitant concomitant treatment ог а therapy which ended less than 7 days before baseline with corticosteroids, diuretics, anticoagulative agents, platelet aggregation inhibitors and systemic/topical use of anti-inflammatory agents, other preparations for veins and analgesics;
* known intolerance against the active ог the inactive ingredients of the study medication (especially lactose);
* pregnancy
* lactation,
* known alcohol or drug abuse
* participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1996-09; Primary Completion 1997-06 (Actual); Study Completion 1997-06 (Actual)

PRIMARY OUTCOMES:
Difference of pain at rest between values day 0 (baseline) and day 7 | Change day 0 until day 7
  Patients were asked to evaluate resting pain on day 0 (baseline) as well as day 7 on a 10-cm VAS (Visual Analogue Scale), with the left end (0 cm) indicating "no pain" and the right end (10 cm) "unbearable pain". The distance from the left end was recorded.
Responders | day 14
  Number of responders (pain value smaller or equal to 1 cm on visual analogue scale for pain (VAS, eft end (0 cm) indicating "no pain" and the right end (10 cm) "unbearable pain") on day 14

OTHER OUTCOMES:
Pain under Pressure | 0, 4, 7, 14 days
  Meyer's pressure points at the lateral side of the tibia and Krieger's pressure point in the popliteal space, 4-point rating scale ranging from 0 (no pain) to 3 (severe pain)
Symptoms | 0, 4, 7, 14 days
  skin redness, hyperthermia, palpable/visible phlebitic cords, heaviness, tenseness
Sum Score of Symptoms | 0, 4, 7, 14 days
  Sum score of all described symptoms (skin redness, hyperthermia, palpable/visible phlebitic cords, heaviness, tenseness)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Baumueller, MD, Principal Investigator — Private Practice; Gerhard Stauder, Dr, Study Director — Mucos Pharma GmbH & Co. KG (EX)
Locations (1):
- Dr. Baumueller, Fano, Italy

IPD SHARING:
Plan to Share IPD: No